CLINICAL TRIAL: NCT00213473
Title: Prospective Clinical and Biological Follow-up of Acquired Haemophilia : SACHA Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2001/001/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Acquired Haemophilia; Register
Keywords: acquired haemophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
the aims of SACHA study was to appreciate prevalence, evolution and follow-up, treatment response of patients with acquired hemophilia with biological and clinical data. Inclusion criteria were factor VIIIc below 30% associated with presence of Facgteur VIII inhibitor (titer > 1 u Bethesda. Clinical and biologival data were obtained at Day 0 (as soon as possible and at 1, 3, 6 and 12 months.Informations were notified to co-investigators with the help of two french medical society (Internal medicine, french haemostasis and thrombosis society.

ELIGIBILITY:
Inclusion Criteria:

* Factor VIIIc < 30% and Factor VIII inhibitor > 1 u Bethesda

Exclusion Criteria:

* absence and signed consent, haemophilia A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with Acquired haemophilia
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2001-06; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Herve LEVESQUE, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- University Hospital of Rouen, Rouen, France

REFERENCES:
- [Derived] Wootla B, Christophe OD, Mahendra A, Dimitrov JD, Repesse Y, Ollivier V, Friboulet A, Borel-Derlon A, Levesque H, Borg JY, Andre S, Bayry J, Calvez T, Kaveri SV, Lacroix-Desmazes S. Proteolytic antibodies activate factor IX in patients with acquired hemophilia. Blood. 2011 Feb 17;117(7):2257-64. doi: 10.1182/blood-2010-07-296103. Epub 2010 Dec 3. PMID 21131590